CLINICAL TRIAL: NCT06754943
Title: A Randomized, Open-label, Single Dose, 2x4 Replicate Crossover Study to Evaluate the Safety and Pharmacokinetic Characteristics After Co-administration of JW0104 and C2402 and Administration of JW0105 in Healthy Volunteers
Brief Title: To Evaluate the Safety and PK Characteristics After Co-administration of JW0104 and C2402 and Administration of JW0105
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JW24102
Record Dates: First submitted 2024-12-10; First posted 2025-01-01 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Healthy
MeSH Terms: interventions — Sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Other): * Treatment A: Co-administration of 1 tablet of JW0104 and 1 tablet of C2402
  * Treatment B: Administration alone of 1 tablet of JW0105
  Interventions: Drug: Treatment A_Period 1; Drug: Treatment B_Period 2; Drug: Treatment A_Period 3; Drug: Treatment B_Period 4
- Group 2 (Other): * Treatment A: Co-administration of 1 tablet of JW0104 and 1 tablet of C2402
  * Treatment B: Administration alone of 1 tablet of JW0105
  Interventions: Drug: Treatment B_Period 1; Drug: Treatment A_Period 2; Drug: Treatment B_Period 3; Drug: Treatment A_Period 4

INTERVENTIONS:
Drug: Treatment A_Period 1 — * Co-administration of 1 tablet of JW0104 and 1 tablet of C2402
  * Wash-out period: 21 days
  * Administration: Treatment A is administered orally with 150 mL of water under fasting conditions
  Other Names: NA (Not Applicable)
  Arms: Group 1
Drug: Treatment B_Period 2 — * Administration alone of 1 tablet of JW0105
  * Wash-out period: 21 days
  * Administration: Treatment B is administered orally with 150 mL of water under fasting conditions
  Other Names: NA (Not Applicable)
  Arms: Group 1
Drug: Treatment A_Period 3 — * Co-administration of 1 tablet of JW0104 and 1 tablet of C2402
  * Wash-out period: 21 days
  * Administration: Treatment A is administered orally with 150 mL of water under fasting conditions
  Other Names: NA (Not Applicable)
  Arms: Group 1
Drug: Treatment B_Period 4 — * Administration alone of 1 tablet of JW0105
  * Wash-out period: 21 days
  * Administration: Treatment B is administered orally with 150 mL of water under fasting conditions
  Other Names: NA (Not Applicable)
  Arms: Group 1
Drug: Treatment B_Period 1 — * Administration alone of 1 tablet of JW0105
  * Wash-out period: 21 days
  * Administration: Treatment B is administered orally with 150 mL of water under fasting conditions
  Other Names: NA (Not Applicable)
  Arms: Group 2
Drug: Treatment A_Period 2 — * Co-administration of 1 tablet of JW0104 and 1 tablet of C2402
  * Wash-out period: 21 days
  * Administration: Treatment A is administered orally with 150 mL of water under fasting conditions
  Other Names: NA (Not Applicable)
  Arms: Group 2
Drug: Treatment B_Period 3 — * Administration alone of 1 tablet of JW0105
  * Wash-out period: 21 days
  * Administration: Treatment B is administered orally with 150 mL of water under fasting conditions
  Other Names: NA (Not Applicable)
  Arms: Group 2
Drug: Treatment A_Period 4 — * Co-administration of 1 tablet of JW0104 and 1 tablet of C2402
  * Wash-out period: 21 days
  * Administration: Treatment A is administered orally with 150 mL of water under fasting conditions
  Other Names: NA (Not Applicable)
  Arms: Group 2

SUMMARY:
The objective is to evaluate the safety and pharmacokinetic characteristics after co-administration of JW0104 and C2402 and administration of JW0105 in healthy volunteers under fasting conditions.

DETAILED DESCRIPTION:
Pharmacokinetic characteristics: Describes the blood concentration statistically by pharmacokinetic blood collection time and treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Subjects does not meet the inclusion Criteria

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
AUCt | Day 1 (0 hour) ~ Day 3 (72 hour) post-dose in period 1, period 2, period 3, and period 4
  Plasma concentrations are measured using a validated LC-MS/MS.
Cmax | Day 1 (0 hour) ~ Day 3 (72 hour) post-dose in period 1, period 2, period 3, and period 4
  Plasma concentrations are measured using a validated LC-MS/MS.

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Dae Kwon, Principal Investigator — Metro Hospital
Locations (1):
- Metro Hospital, Anyang-si, Gyeonni-do, South Korea

IPD SHARING:
Plan to Share IPD: No